CLINICAL TRIAL: NCT01735305
Title: Optimal Antiplatelet Therapy for Chinese Patients With Coronary Artery Disease
Acronym: OPT-CAD
Status: Completed | Type: Observational
Sponsor: Shenyang Northern Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Dr, Shenyang Northern Hospital
Other Study IDs: SYNH-20121113
Record Dates: First submitted 2012-11-12; First posted 2012-11-28 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; antiplatelet therapy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Antiplatelet therapy: patients with coronary artery disease receiving any antiplatelet therapy, without any intervention by the investigators.

SUMMARY:
Antiplatelet therapy is the cornerstone for the prevention of atherothrombosis in patients with coronary artery disease (CAD). However, the efficacy and safety of antiplatelet therapy are varied due to ethnic and/or individual variability. The aim of the OPT-CAD study was to demonstrate contemporary status and outcomes of antiplatelet therapy in Chinese CAD patients, and to explore predictors of ischemic or bleeding events in such cohort.Patients above 18 years old who were diagnosed as CAD and received antiplatelet therapy were prospectively enrolled in this national wide, non-intervention registry. All medications and laboratory tests were physician discretion.

DETAILED DESCRIPTION:
Antiplatelet therapy is the cornerstone for the prevention of atherothrombosis in patients with coronary artery disease (CAD). However, the efficacy and safety of antiplatelet therapy are varied due to ethnic and/or individual variability. The aim of the OPT-CAD study was to demonstrate contemporary status and outcomes of antiplatelet therapy in Chinese CAD patients, and to explore predictors of ischemic or bleeding events in such cohort.Patients above 18 years who were diagnosed as CAD and received antiplatelet therapy were prospectively enrolled in this national wide, non-intervention registry. All medications and laboratory tests were at physician discretion.

ELIGIBILITY:
Inclusion criteria:

1. Clinical diagnosis of coronary heart disease
2. Age >= 18 years old
3. receiving any antiplatelet agents
4. Informed written consent signed

Exclusion Criteria:

1. With severe disease and life expectancy for 6 months or less
2. Difficult to attain follow-up situations judged by researchers (travel, speech or mental disorder, etc.)
3. Taking part in an interventional clinical research

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient of coronary heart disease receiving any antiplatelet therapy
Sampling Method: Non-Probability Sample
Enrollment: 14032 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebral events | 12month
  a composite of all cause death, myocardial infarction, stroke or any revascularization or stroke

SECONDARY OUTCOMES:
all cause death | 12month
Stent thrombosis | 12 month
  by BARC definition
rehospitalization | 12 month
  any rehospitalization for cardiac or noncardiac reasons
any bleeding events | 12 month
  by BARC definition
recurrent angina | 12 month
myocardial infarction | 12 months
stroke | 12 months
any revascularization | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — Shenyang Military Region General Hospital
Locations (107):
- China (107):
  - The first affiliated hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Navy General Hospital, Beijing, Beijing Municipality
  - The 304th Hospital of PLA, Beijing, Beijing Municipality
  - The 306th of PLA, Beijing, Beijing Municipality
  - The Luhe teaching hospital of the Capital Medical University, Beijing, Beijing Municipality
  - The People's Hospital of Beijing University, Beijing, Beijing Municipality
  - Yanshan hospital, Beijing, Beijing Municipality
  - Beijing Fuwai Hospital, Beijin, Beijing Municipality
  - Third Military Medical University Xinqiao Hospital, Chongqing, Chongqing Municipality
  - The 174th Hospital of PLA, Xiamen, Fujian
  - Lanzhou military region general hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou Medical College, Guangdong, Guangdong
  - General hospital of armed police foreces in Guangzhou, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Guangzhou Baiyun district hospital, Guangzhou, Guangdong
  - Guangzhou military region general hospital, Guangzhou, Guangdong
  - Guangzhou Panyu district central hospital, Guangzhou, Guangdong
  - Liwan District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The first hospital of Guangzhou, Guangzhou, Guangdong
  - Shenzhen Longgang center hospital, Shenzhen, Guangdong
  - Zhuhai people's hospital, Zhuhai, Guangdong
  - The 3rd people's hospital of Nanning, Nanning, Guangxi
  - Guizhou provincial people's hospital, Guiyang, Guizhou
  - The 425th of PLA, Sanya, Hainan
  - Affiliated hospital of Hebei University of Engineering, Handan, Hebei
  - The People's Hospital of Tangxian, Renhou, Hebei
  - The people's hospital of Rongcheng, Rongcheng, Hebei
  - Bethune International Peace Hospital, Shijiazhuang, Hebei
  - The 251st of PLA, Zhangjiakou, Hebei
  - Daqing oil field hospital, Daqing, Heilongjiang
  - Heilongjiang provincial hospital, Harbin, Heilongjiang
  - The 211st of PLA, Harbin, Heilongjiang
  - The third affiliated hospital of Qiqihar Medical University, Qiqihar, Heilongjiang
  - The People's Hospital of Hebi, Hebi, Henan
  - The 152nd Hospital of PLA, Pingdingshan, Henan
  - The People's Hospital of Zhecheng County, Zhecheng Chengguanzhen, Henan
  - The First Hospital of Organization Directly Under Henan Province, Zhengzhou, Henan
  - Wuhan Asia heart hospital, Wuhan, Hubei
  - The first hospital of Changshan, Changshan, Hunan
  - The general hospital of Xilingol League, Mositai, Inner Mongolia
  - The first hospital of Nanjing, Nanjing, Jiangsu
  - The central hospital of Nantong, Nantong, Jiangsu
  - The Affiliated Hospital of Jinggangshan University, Ji’an, Jiangxi
  - Central Hospital of Changchun, Changchun, Jilin
  - The affiliated hospital to Changchun University of Chinese Medicine, Changchun, Jilin
  - The China-Japan union hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Jilin University, Changchun, Jilin
  - The Second Affiliated Hospital of Jilin University, Changchun, Jilin
  - The 222nd of PLA, Jilin, Jilin
  - Meihekou central hospital, Meihekou, Jilin
  - Siping first people's hospital, Siping, Jilin
  - The 206th of PLA, Tonghua, Jilin
  - The people's hospital of Tonghua, Tonghua, Jilin
  - Tonghua central hospital, Tonghua, Jilin
  - Anshan central hospital, Anshan, Liaoning
  - Anshan hospital affiliated of China Medical University, Anshan, Liaoning
  - The first affiliated hospital of Liaoning Medical University, Anshan, Liaoning
  - The people's hospital of Xiuyan, Anshan, Liaoning
  - The third hospital of Anshan, Anshan, Liaoning
  - Dalian municipal central hospital affiliated of Dalian Medical University, Dalian, Liaoning
  - The 210th Hospital of PLA, Dalian, Liaoning
  - Zhongshan Hospital Affiliated to Dalian University, Dalian, Liaoning
  - The 230th of PLA, Dandong, Liaoning
  - The people's hospital of Dandong, Dandong, Liaoning
  - Central Hospital affiliated to Shenyang Medical College, Fengtian, Liaoning
  - Fushun central hospital, Fushun, Liaoning
  - The 7th hospital of China Medical University, Fushun, Liaoning
  - The Second Affiliated and gynecology and obstetirs hospital of Fuxin city, Fuxin, Liaoning
  - The people's hospital of Haicheng, Haicheng, Liaoning
  - The 205th of PLA, Jinzhou, Liaoning
  - The third affiliated hospital of Liaoning medical College, Jinzhou, Liaoning
  - Central hospital of Liaoyang, Liaoyang, Liaoning
  - Liaoyang Chemical General Hospital, Liaoyang, Liaoning
  - The 201th Hospital of PLA, Liaoyang, Liaoning
  - The 2nd people's hospital of Liaoyang, Liaoyang, Liaoning
  - Jinqiu Hospital, Shenyang, Liaoning
  - Liaoning northern hospital, Shenyang, Liaoning
  - Shenyang the forth hospital of people, Shenyang, Liaoning
  - The 202nd Hospital of PLA, Shenyang, Liaoning
  - The 242nd of PLA, Shenyang, Liaoning
  - The 245th of PLA, Shenyang, Liaoning
  - The 463rd Hospital of PLA, Shenyang, Liaoning
  - The First Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The first people's hospital of Shenyang, Shenyang, Liaoning
  - The Forth affiliated hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The Second Affiliated Hospital of Shenyang Medical College, Shenyang, Liaoning
  - The Third Affiliated Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Traditional Chinese Medicine hospital of Shenyang, Shenyang, Liaoning
  - Yingkou Development Zone Hospital, Yingkou, Liaoning
  - General hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The people's hospital of Huzhu, Huzhu, Qinghai
  - Tangdu hospital, Xi'an, Shaanxi
  - Jinan military general hospital, Jinan, Shandong
  - Jiaozhou central hospital, Qingdao, Shandong
  - Wanjie Hospital, Zibo, Shandong
  - Eastern hospital in Shanghai, Shanghai, Shanghai Municipality
  - Yuncheng central hospital, Yuncheng, Shanxi
  - Sichuan military general hospital, Chengdu, Sichuan
  - Armed police foreces'hospital of Tianjin, Tianjin, Tianjin Municipality
  - The 254th of PLA, Tianjin, Tianjin Municipality
  - Xizang military general hospital, Lhasa, Tibet
  - The 11st of PLA, Huiyuan, Xinjiang
  - General hospital of Wulumuqi, Ürümqi, Xinjiang
  - The Chest Hospital of Xinjiang Uyghur Autonomous Region, Ürümqi, Xinjiang
  - The 4th public hospital of Honghe, Yisa, Yunnan
  - Hangzhou first people's hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Ma S, Jiang Z, Qiu M, Li Z, Bian L, Li Y, Han Y. Dual Antiplatelet Therapy Duration in Medically Managed Acute Coronary Syndrome Patients: Sub-Analysis of the OPT-CAD Study. Adv Ther. 2020 Jul;37(7):3150-3161. doi: 10.1007/s12325-020-01376-0. Epub 2020 May 16. PMID 32418142
- [Derived] Feng YQ, He XY, Song FE, Chen JY. Association between Contrast Media Volume and 1-Year Clinical Outcomes in Patients Undergoing Coronary Angiography. Chin Med J (Engl). 2018 Oct 20;131(20):2424-2432. doi: 10.4103/0366-6999.243563. PMID 30334527